CLINICAL TRIAL: NCT06575608
Title: Estimation of VO2Max Using Smartphone Application in Elderly: Validation Study
Brief Title: Estimation of VO2Max Using Smartphone Application
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Abd El-satar Mohamed Said, principal investigator, Cairo University
Other Study IDs: P.T.REC/012/004899
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-08

CONDITIONS: Assessmet of VO2max in Elderly
Keywords: VO2MAX; Smartphone application; Elderly; cardiorespiratory fitness (CRF)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- direct VO2max test group: Group A (n-26) will perform a direct VO2max test on the treadmill and vo2max will be calculated by the cardiopulmonary exercise testing (CPX) device Spirometry Medisoft Ergocart professional.
- 1-mile walk test group: Group B (n-26) will perform the 1 mile walk test and VO2 max will be calculated by the smartphone application VO2max calculator

SUMMARY:
The aim of this observational study Is to examine the validity of the Smartphone application (VO2max calculator) in calculating VO2max in elderly population.

Research hypotheses:

this study will test the following null hypothesis: (Vo2max calculator) application will not have criterion validity in estimating VO2max values in the elderly population.

Research question:

Is the Smartphone application (VO2max calculator) considered a valid tool for estimating accurate values of VO2max in the elderly population in comparison to the golden standard method?

DETAILED DESCRIPTION:
Although maximal oxygen consumption (VO2max) is growing in evidence as a powerful indicator of several health conditions it's rarely used in clinical practice due to the high expense, requirement of specialized equipment, and related risks of maximal exertion. So, we aim to develop a simpler method for estimating VO2max using modern smartphone technologies.

Method: participants of this study will be divided into 2 equal groups. The first group will perform a gold standard treadmill-based VO2max measurement and the other group will perform a smartphone based 1-mile walk test for VO2max estimation.

ELIGIBILITY:
Inclusion Criteria:

* Elderly subjects aged from (65 to 75) years.
* BMI 18.5-29.9 kg/m2
* Answer (NO) to all of the questions in the Physical activity readiness questionnaire (PAR-Q)
* Do not have any absolute or relative contraindications for exercise testing according to the American Heart Association (AHA) statement.

Exclusion Criteria:

* Recent surgical conditions.
* Skeletal deformities.
* Blood pressure regulating medication intake.
* Any respiratory disorders.
* Back, hip, knee or ankle pain within last month.
* Any neurological or psychiatric conditions.
* Implanted pacemaker.
* Anemic patients.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: (52) Male and female participants will be recruited from the out clinic customers, and workers at the faculty of physical therapy Delta University at ELmansoura governorate.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
maximum oxygen consumption (VO2MAX) | at the peak of exercise (peak VO2) over the final 30 seconds of exercise
  The greatest amount of oxygen a person can take in from inspired air while performing dynamic exercise involving a large part of total muscle mass.

SECONDARY OUTCOMES:
Heart rate (HR) | at baseline one shot
  the number of times your heart beats per minute.
The Borg rating of perceived exertion (RPE) scale | at baseline one shot
  It is a subjective scale for estimating effort and exertion, breathlessness, and fatigue during physical work.